CLINICAL TRIAL: NCT03064698
Title: Uterine Artery Doppler Changes From the Second Trimester of Pregnancy to the Postpartum Period in a Group of High Risk Women
Brief Title: Uterine Artery Doppler Changes
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 16-035
Record Dates: First submitted 2017-02-13; First posted 2017-02-27 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Uterine Artery Flow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal second trimester Doppler: This group consists of women who had normal doppler ultrasound results at second trimester
  Interventions: Other: Post-partum Doppler ultrasound
- Abnormal second trimester Doppler: This group consists of women who had abnormal doppler ultrasound results at second trimester
  Interventions: Other: Post-partum Doppler ultrasound

INTERVENTIONS:
Other: Post-partum Doppler ultrasound — Participants will undergo one uterine artery Doppler ultrasound at 6 weeks post-partum.

SUMMARY:
In uncomplicated pregnancies, the uterine spiral arteries undergo a series of structural changes that result in a low resistance in the uterine arteries as pregnancy progresses.

In many pregnancies complicated with preeclampsia, growth restriction and other placental related complication, the described change does not occur. In pregnancies at high risk for placental complications, doppler measurement of Uterine artery flow has been shown to be a reliable predictor of complications.

Postpartum there is a reversal of vascular changes seen in normal pregnancies. It is unclear if there is a full reversal of these changes in complicated pregnancies with abnormal flow during pregnancy.

The investigators hypothesize that Doppler uterine artery measurements after complicated pregnancies will show some abnormality compared to doppler measurements following uncomplicated pregnancies.

DETAILED DESCRIPTION:
The postpartum reversal of pregnancy-related changes in uterine artery (UA) flow is not well documented.

While long-term vascular changes have been noted in women with prior preeclampsia (PE), and in a dose- dependent manner, long-term changes to UA vascular resistance following PE have not been analyzed. Moreover, regardless of whether they experienced PE or intrauterine growth restriction (IUGR), it is not known if women with elevated UA pulsatility index (PI) in mid-pregnancy have higher UA well after pregnancy, compared to women whose UA PI was normal in mid-pregnancy.

The investigators propose to evaluate if UA flow remains abnormally high postpartum in women who had elevated UA flow mid-pregnancy, compared to women whose UA flow was normal in mid-pregnancy.

This is an observational prospective study. The study recruits women that have recently delivered and have undergone a Uterine Doppler ultra sound (US) during the second trimester of their pregnancy. Eligible women will undergo one post-partum ultrasound examination.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent UA Doppler assessment at 18-22 weeks gestation.
* Viable singleton pregnancy at the time of UA Doppler assessment at 18-22 weeks gestation.
* Is at least 6 weeks postpartum following a livebirth of the aforementioned pregnancy
* Not pregnant at time of post-partum UA Doppler assessment

Exclusion Criteria:

* Women will be excluded if they do not meet the above criteria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Women with singleton pregnancies.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in uterine artery flow | 2nd trimester (between 13 to 22 weeks gestation) and 6 weeks post-partum
  Uterine artery flow measurements during pregnancy and after, as measured by Doppler ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Howard Berger, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No